CLINICAL TRIAL: NCT03372915
Title: Testing an Inhibitory Learning Model of Extinction in Exposure-Based Anxiety Treatment for Youth: Feasibility, Acceptability, and Efficacy
Brief Title: Test of an Inhibitory Learning Model of Extinction in Treatment of Anxious Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17-2040
Record Dates: First submitted 2017-11-28; First posted 2017-12-14 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Anxiety Disorders
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Exposure (Active Comparator): This arm will receive exposure therapy conducted according to standard care practices.
  Interventions: Behavioral: Standard Exposure
- Exposure + Inhibitory Learning (Experimental): This arm will receive exposure therapy conducted according to principles of inhibitory learning.
  Interventions: Behavioral: Exposure + Inhibitory Learning

INTERVENTIONS:
Behavioral: Standard Exposure — Exposure therapy conducted according to standard clinical care practices
  Arms: Standard Exposure
Behavioral: Exposure + Inhibitory Learning — Exposure therapy conducted according to practice recommendations based derived from research on inhibitory learning theories of fear extinction
  Arms: Exposure + Inhibitory Learning

SUMMARY:
Recently, basic research conducted in adults has revealed that fear extinction, or the weakening of a learned fear response, may be best explained by principles of "inhibitory learning." New guidelines for the clinical practice of exposure therapy for anxiety disorders have arisen from research on inhibitory learning, but these guidelines have not yet been empirically tested in youth with anxiety disorders. The overall goal of this research is to investigate the acceptability, feasibility, and efficacy of conducting exposure therapy for anxiety disorders in youth according to clinical guidelines developed from basic research on inhibitory learning principles, using a pilot randomized controlled trial design.

DETAILED DESCRIPTION:
Exposure therapy-which involves repeatedly exposing individuals to feared situations to change their fear responses to and beliefs about those situations--has been a mainstay of treatments for anxiety disorders since it was developed in the 1950s. Today, exposure therapy is the most commonly-occurring treatment technique included in well-supported treatments for anxiety disorders, and meta-analyses have indicated that exposure is more strongly associated with treatment gains in anxious youth compared to non-behavioral interventions. Despite its effectiveness, approximately 40% of anxious youth fail to achieve clinically significant benefit from exposure therapy. This indicates that further research is needed regarding strategies for optimizing exposure therapy so that it is effective for a greater proportion of youth.

There is clearly a need to optimize exposure therapy for youth, but at the same time very little empirical data exists regarding how exposure works or the best way to conduct exposures. Common wisdom about exposure, based on emotional processing theory, dictates that exposure works by breaking and eliminating conditioned fear responses through a process called habituation. This viewpoint dictates that exposure should be conducted until habituation occurs (i.e., until a physiological fear response reduces by at least 50%), and that habituation both during and between exposure sessions is necessary for improvement. As exposure therapy has evolved, other common practices have emerged that lack clear evidence supporting their efficacy. For example, it is common clinical practice to encourage youth to challenge their thoughts about a feared situation before and during an exposure (i.e., cognitive restructuring), even though clear evidence does not exist to support this practice. Additionally, it is common for clinicians to create a "fear ladder" or "hierarchy" with patients before beginning exposures. This hierarchy typically takes the form of a rank-ordered list of exposures or feared stimuli from least to most difficult, and clinicians move up this list systematically from the easiest to most difficult items during treatment. Again, there is little clear evidence to support this practice.

More recent research on fear extinction indicates that exposure therapy does not cause threat associations to disappear but rather leads to the formation of non-threat (i.e., inhibitory) associations that compete with and weaken older threat associations. The goal of exposure therapy, according to this model, is to strengthen these non-threat associations and weaken threat associations. Research on inhibitory learning has turned many of the long-standing exposure practices discussed in the previous paragraph on their head by providing new guidelines for optimizing exposure therapy. Many of these new guidelines differ significantly from common clinical practices and are designed to maximize learning of inhibitory associations. These guidelines are as follows:

1. Design exposures that maximally violate a patient's expectations about how bad an outcome would be or how often it will occur. In clinical practice, an exposure that maximally violates expectancies is one that is terminated not when fear habituates or reduces by a certain amount (e.g., "What is your fear rating?") but rather when the patient's expectancy of a bad outcome is significantly reduced. (e.g., "What do you think the chances are that X will happen?).
2. Do not instruct patients to change their thinking about a feared situation before or during and exposure. The principle of maximum violation of expectancies dictates that participants should not be encouraged to use cognitive reappraisal (e.g., strategies for thinking more realistically or accurately) during an exposure, as such strategies reduce the expectation that a negative outcome will occur and thus prevent maximum violation of expectancy.
3. Introduce variability of stimuli into exposure tasks by moving up and down a fear ladder randomly. Inhibitory learning theory suggests that clinicians should frequently vary the difficulty of exposure to stimuli to create a consistently high level of emotion, which has been associated with superior extinction learning. This guideline means that, instead of moving up a fear hierarchy or ladder in a systematic way from least to most difficult over time, and moving on to more difficult items after habituation to easier ones has occurred, clinicians should design exposures that will allow patients to achieve variable but generally high levels of fear or anxiety over the full course of an exposure.

In this study, the investigators plan to test these clinical practice guidelines derived from inhibitory learning against standard exposure practice. A few studies have empirically tested these and/or other clinical practice guidelines established based on inhibitory learning in clinical adult samples. However, no known studies have yet empirically tested the efficacy of an inhibitory learning approach to exposure therapy in youth with anxiety or other emotional disorders, nor have any known studies tested the acceptability or feasibility of such an approach. Therefore, in this study the investigators propose to conduct a small-scale, pilot randomized controlled trial (RCT) examining the feasibility, acceptability, and relative efficacy of applying an inhibitory learning approach to exposure in youth. Up to 20 youth will be randomized to one of two groups-standard exposure (SE) or exposure conducting according to inhibitory learning principles (E + IL). Given the small n for this study, the primary goal will be to assess feasibility and acceptability of an inhibitory learning approach to exposure, while establishing the efficacy of this approach relative to SE is exploratory. This study, along with planned larger-scale RCTs to follow, will help to inform clinical care guidelines for best practice of exposure therapy with anxious youth.

ELIGIBILITY:
Inclusion Criteria:

1. Primary or secondary diagnosis of an anxiety disorder
2. Ability of both child and caregiver to read and understand English
3. Ability of child and at least one caregiver to attend weekly sessions

Exclusion Criteria:

1. Diagnosis of autism spectrum disorder, intellectual development disorder, or limited cognitive functioning (i.e., documented Intelligence Quotient [IQ]<80).
2. Diagnosis of a psychotic disorder or bipolar disorder
3. Severe and current suicidal ideation, history of suicide attempt in past six months, or frequent and persistent self-injurious behavior
4. Diagnosis of a substance use disorder or significant, recent substance use
5. Any youth receiving concurrent individual therapy will also be excluded from the study.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2018-01-31 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Change in Percentage of Exposure Refusals (Feasibility Measure) | Treatment weeks 5, 6, 7, and 8
  Therapists will record the percentage of exposures the patient refused to complete during the session.
Change in Latency to Initiating Exposure (Feasibility Measure) | Treatment weeks 5, 6, 7, 8
  Therapist will record the average amount of time the patient delayed before initiating each exposure in session
Early Treatment Termination (Feasibility Measure) | Measure will be collected following the patient's termination from treatment
  Information will be collected regarding whether the patient terminated treatment early (before session 9)
Change in Homework Completion (Feasibility Measure) | Treatment weeks 6, 7, 8, and 9
  Therapist will record the number of exposure sessions for which the patient completed homework
Client Satisfaction Questionnaire-8 (CSQ-8) | Week 9 (End of Treatment)
  8-item measure of patient satisfaction with treatment. The measure is rated on a four-point scale, with possible scores ranging from 8-32.

SECONDARY OUTCOMES:
Change in Distress Tolerance Scale--Child (DTS-C) | Treatment Week 1, Week 5, and Week 9 (End of Treatment)
  A 15-item self-report measure of difficulties managing distress and related emotions. The measure is rated on a 5-point scale, with possible scores ranging from 15 to 65. Higher scores indicate greater ability to tolerate distress.
Change in Child Avoidance Measure, Self and Parent Report (CAMS/P) | Treatment Week 1, Week 5, and Week 9 (End of Treatment)
  The CAMS/P are 8-item child- and parent-report (respectively) measures of behavioral avoidance. The measure is rated on a 4-point scale, with possible scores ranging from 0 to 24. Higher scores indicate greater behavioral avoidance.
Change in Avoidance and Fusion Questionnaire--Youth (AFQ-Y) | Treatment Week 1, Week 5, and Week 9 (End of Treatment)
  A 17-item self-report measure of experiential avoidance and cognitive fusion. The measure is rated on a 4-point scale, with possible scores ranging from 0 to 68. Higher scores indicate greater cognitive fusion and experiential avoidance.
Change in Parent Acceptance and Action Questionnaire (PAAQ) | Treatment Week 1, Week 5, and Week 9 (End of Treatment)
  A 15-item measure of parent experiential avoidance, or parental actions intended to control the form and frequency of their child's emotional experiences. Items are rated on a 7-point scale, with possible scores ranging from 17 to 105. Higher scores indicate less parental experiential avoidance and less effort to control child emotional experiences.
Change in Screen for Child Anxiety Related Disorders (SCARED), Self and Parent Report | Treatment Week 1, Week 5, Week 6, Week 7, Week 8, and Week 9 (End of Treatment)
  A 41-item child- and parent-report measure assessing symptoms of anxiety in youth ages 7 to 19. Items are rated on a 3-point scale, with scores ranging from 0 to 82. Higher scores indicate greater anxiety symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Hawks, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Arch, J. J., & Abramowitz, J. S. (2015). Exposure therapy for obsessive-compulsive disorder: An optimizing inhibitory learning approach. Journal of Obsessive-Compulsive and Related Disorders, 6, 174-182.
- [Background] Birmaher B, Khetarpal S, Brent D, Cully M, Balach L, Kaufman J, Neer SM. The Screen for Child Anxiety Related Emotional Disorders (SCARED): scale construction and psychometric characteristics. J Am Acad Child Adolesc Psychiatry. 1997 Apr;36(4):545-53. doi: 10.1097/00004583-199704000-00018. PMID 9100430
- [Background] Cheron DM, Ehrenreich JT, Pincus DB. Assessment of parental experiential avoidance in a clinical sample of children with anxiety disorders. Child Psychiatry Hum Dev. 2009 Sep;40(3):383-403. doi: 10.1007/s10578-009-0135-z. Epub 2009 Mar 12. PMID 19280337
- [Background] Craske MG, Kircanski K, Zelikowsky M, Mystkowski J, Chowdhury N, Baker A. Optimizing inhibitory learning during exposure therapy. Behav Res Ther. 2008 Jan;46(1):5-27. doi: 10.1016/j.brat.2007.10.003. Epub 2007 Oct 7. PMID 18005936
- [Background] Craske MG, Treanor M, Conway CC, Zbozinek T, Vervliet B. Maximizing exposure therapy: an inhibitory learning approach. Behav Res Ther. 2014 Jul;58:10-23. doi: 10.1016/j.brat.2014.04.006. Epub 2014 May 9. PMID 24864005
- [Background] Deacon B, Kemp JJ, Dixon LJ, Sy JT, Farrell NR, Zhang AR. Maximizing the efficacy of interoceptive exposure by optimizing inhibitory learning: a randomized controlled trial. Behav Res Ther. 2013 Sep;51(9):588-96. doi: 10.1016/j.brat.2013.06.006. Epub 2013 Jul 6. PMID 23872701
- [Background] Ehrenreich-May, J., Kennedy, S. M., Sherman, J., Bilek, E. L., Buzzella, B., Bennett, S., & Barlow, D. H. (In press). Unified protocols for transdiagnostic treatment of emotional disorders in children and adolescents. New York: Oxford University Press.
- [Background] Foa EB, Kozak MJ. Emotional processing of fear: exposure to corrective information. Psychol Bull. 1986 Jan;99(1):20-35. No abstract available. PMID 2871574
- [Background] Greco LA, Lambert W, Baer RA. Psychological inflexibility in childhood and adolescence: development and evaluation of the Avoidance and Fusion Questionnaire for Youth. Psychol Assess. 2008 Jun;20(2):93-102. doi: 10.1037/1040-3590.20.2.93. PMID 18557686
- [Background] Higa-McMillan CK, Francis SE, Rith-Najarian L, Chorpita BF. Evidence Base Update: 50 Years of Research on Treatment for Child and Adolescent Anxiety. J Clin Child Adolesc Psychol. 2016;45(2):91-113. doi: 10.1080/15374416.2015.1046177. Epub 2015 Jun 18. PMID 26087438
- [Background] Larsen DL, Attkisson CC, Hargreaves WA, Nguyen TD. Assessment of client/patient satisfaction: development of a general scale. Eval Program Plann. 1979;2(3):197-207. doi: 10.1016/0149-7189(79)90094-6. No abstract available. PMID 10245370
- [Background] Milad MR, Pitman RK, Ellis CB, Gold AL, Shin LM, Lasko NB, Zeidan MA, Handwerger K, Orr SP, Rauch SL. Neurobiological basis of failure to recall extinction memory in posttraumatic stress disorder. Biol Psychiatry. 2009 Dec 15;66(12):1075-82. doi: 10.1016/j.biopsych.2009.06.026. Epub 2009 Sep 12. PMID 19748076
- [Background] Muris, P., Merckelbach, H., van Brakel, A., Mayer, B., & van Dongen, L. (1998). The Screen for Child Anxiety Related Emotional Disorders (SCARED): Relationship with anxiety and depression in normal children. Personality and Individual Differences, 24(4), 451-456.
- [Background] Shin LM, Liberzon I. The neurocircuitry of fear, stress, and anxiety disorders. Neuropsychopharmacology. 2010 Jan;35(1):169-91. doi: 10.1038/npp.2009.83. PMID 19625997
- [Background] Simons, J. S., & Gaher, R. M. (2005). The Distress Tolerance Scale: Development and validation of a self-report measure. Motivation and Emotion, 29(2), 83-102.
- [Background] Whiteside SP, Ale CM, Young B, Dammann JE, Tiede MS, Biggs BK. The feasibility of improving CBT for childhood anxiety disorders through a dismantling study. Behav Res Ther. 2015 Oct;73:83-9. doi: 10.1016/j.brat.2015.07.011. Epub 2015 Jul 29. PMID 26275761
- [Background] Whiteside SP, Gryczkowski M, Ale CM, Brown-Jacobsen AM, McCarthy DM. Development of child- and parent-report measures of behavioral avoidance related to childhood anxiety disorders. Behav Ther. 2013 Jun;44(2):325-37. doi: 10.1016/j.beth.2013.02.006. Epub 2013 Mar 4. PMID 23611081